CLINICAL TRIAL: NCT00654953
Title: Sertraline Augmented With GABA Agents for Cocaine Dependence
Brief Title: Clinical Efficacy of Sertraline Augmented With Gabapentin in Depressed, Recently Abstinent Cocaine-dependent Humans
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Alison Oliveto Beaudoin, UAMS
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P50DA018197 (NIH); P50DA018197 (NIH); DPMCDA
Record Dates: First submitted 2008-04-04; First posted 2008-04-09 (Estimated); Results first posted 2011-04-25 (Estimated); Last update posted 2011-04-25 (Estimated); Status verified 2011-03

CONDITIONS: Cocaine Dependence; Depressive Symptoms
Keywords: cocaine dependence; depressive symptoms; relapse; sertraline; gabapentin
MeSH Terms: conditions — Cocaine-Related Disorders; Depression; Recurrence | interventions — Sertraline; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Placebo Comparator): Placebo capsules
  Interventions: Drug: Placebo
- 2 (Experimental): sertraline (200 mg/day)
  Interventions: Drug: sertraline; Drug: Placebo
- 3 (Experimental): sertraline (200 mg/day) plus gabapentin (1,200 mg/day)
  Interventions: Drug: sertraline; Drug: gabapentin

INTERVENTIONS:
Drug: sertraline — Sertraline hydrochloride (200 mg/day) will be administered once daily. While subjects are at RCA-NLR they initially receive 50 mg/day of sertraline. This dose is gradually increased over a 3-week period until subjects receive 200 mg. When subjects are transferred to the outpatient program, they will be administered capsules once weekly, with take-home doses given in blister packs to take once a day for the rest of the week.
  Arms: 2; 3
Drug: Placebo — Placebo (cellulose or lactose) administered twice per day for 12 weeks.
  Arms: 1; 2
Drug: gabapentin — Gabapentin (Neurontin; Parke-Davis; 1200 mg/day) will be administered twice daily. Initially, patients will receive 200 mg twice daily on days 1-5, 400 mg twice daily on days 6-10, then 600 mg twice daily on days 11 on. Subjects are then maintained on this dose for the duration of the trial, unless side-effects are too severe, in which case the dose of gabapentin is decreased to no less 800 mg/day. If symptoms persist, subjects' participation would then be terminated.
  Arms: 3

SUMMARY:
To examine the clinical efficacy of sertraline (200 mg/day) alone or sertraline in combination with gabapentin. The purpose of this study is to examine whether the antidepressant sertraline alone or combined with gabapentin delays time to relapse relative to placebo in recently abstinent cocaine-dependent volunteers who are also depressed. In addition, whether depressive symptoms or genetic factors influence treatment response to the study medications will be examined. Our hypothesis is that those on combined sertraline-gabapentin will show a longer period of abstinence than those on sertraline alone or placebo.

DETAILED DESCRIPTION:
Subjects enrolled in this 12-wk, double blind, randomized, placebo-controlled, clinical trial are admitted to a residential facility in North Little Rock (RCA-NLR) and randomized by depressive symptom severity to receive one of the following: sertraline alone (200 mg/day), sertraline (200 mg/day) plus gabapentin (1200 mg/day), or placebo. Subjects are expected to participate in the Substance Abuse Day Treatment Program while residing on the RCA-NLR and being inducted onto the maintenance dose of study medication (weeks 1-2). When participants transfer to the Outpatient Treatment Research Unit (TRU) at the start of their third week, they will continue to receive study medications or placebo (weeks 3-12) and they will be expected to participate in weekly individual cognitive behavioral therapy. Supervised urines and vital signs will be obtained thrice weekly; self-reported adverse effects, mood and drug use self-reports will be obtained once weekly. At the end of 12 weeks, participants will be tapered off the study medication over a five-day period, discharged from the study, and referred to an appropriate treatment or treatment/research program in the community if they are interested.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* not currently enrolled in a treatment program
* subjects must have a history of cocaine use, with street cocaine use by history being a minimum of 1 gram during the preceding 3 months
* subjects must meet DSM-IV criteria for cocaine dependence as assessed by the substance abuse section of the Structured Clinical Interview for DSM-IV (SCID and SCID-SAC)
* subjects must have laboratory confirmation of recent cocaine use (positive urine for cocaine or benzoylecgonine) during the month prior to study entry
* subjects must score at least 15 on the Hamilton Depression Scale
* women of childbearing age must have a negative pregnancy test to enroll in this study and must agree to monthly pregnancy testing

Exclusion Criteria:

* current diagnosis of other drug or alcohol physical dependence (other than cocaine or tobacco)
* ill health (e.g., major cardiovascular, renal, endocrine, hepatic disorder)
* history of schizophrenia, or bipolar type I disorder
* present or recent use of over-the-counter or prescription psychoactive drug or drug(s) that would be expected to have major interaction with drug to be tested
* medical contraindication to receiving study medications (e.g., for sertraline, use of monoamine oxidase inhibitor within last two weeks; significant history of seizures; significant history of head trauma or serious neurological disorders)
* current suicidality or psychosis
* Liver function tests (i.e., liver enzymes) greater than three times normal levels
* pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2006-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, PhD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 143 cocaine-using volunteers gave informed consent between 12/15/2005 and 4/8/2009. Consenting occurred at either the UAMS substance abuse treatment clinic, treatment research unit or center for addiction research at the UAMS Psychiatric Research Institute. Of these, 105 eligible participants were enrolled into the study proper.
Pre-assignment Details: Of the 143 screened, 42 failed randomization/screening procedures and so were not randomized to receive study medication or placebo.
Groups:
- Placebo Group: Placebo capsules
- Active Group: Sertraline Alone: sertraline (200 mg/day)
- Active Group: Sertraline Plus Gabapentin: sertraline (200 mg/day) plus gabapentin (1,200 mg/day)
Period: Overall Study
Arm/Group | Placebo Group | Active Group: Sertraline Alone | Active Group: Sertraline Plus Gabapentin
Started | 36 | 36 | 30
Completed | 6 | 8 | 8
Not Completed | 30 | 28 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Active Group: Sertraline Alone | Active Group: Sertraline Plus Gabapentin | Total
Number analyzed (Participants) | 36 | 36 | 30 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 36 | 36 | 30 | 102
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 38.74 (6.32) | 39.78 (8.36) | 39.40 (7.81) | 39.31 (7.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 6 | 28
  Male | 24 | 26 | 24 | 74
Region of Enrollment [Number; unit: participants]
  United States | 36 | 36 | 30 | 102

OUTCOME MEASURES:

1. Primary Outcome: Urine Toxicology Screens for the Presence of Cocaine/Cocaine Metabolites
Description: Thrice-weekly urine samples were analyzed for the presence of cocaine/cocaine metabolite. Days to Relapse was defined as time to the second of two urine results consecutively positive for cocaine.
Time Frame: 70 days
Population: Participants who completed the two-week residential stay and had 2 urine samples consecutively positive for cocaine were included in the analysis.
Measure: Mean (Standard Deviation); unit: Days to relapse (two consec coc+ urines)
Units Other Than Participants: urine samples
Arm/Group | Placebo | Sertraline | Sertraline Plus Gabapentin
Number analyzed (Participants) | 14 | 8 | 11
Number analyzed (urine samples) | 30 | 30 | 30
Days to relapse (two consec coc+ urines) | 19.93 (12.16) | 23.38 (17.82) | 17.27 (14.49)
Statistical Analysis 1: Comparison: Placebo vs Sertraline vs Sertraline Plus Gabapentin; The analysis tested the null hypothesis of no difference among groups in terms of the # of days to relapse (first two conseqcutively positive urines) using ANOVA; Test type: Superiority or Other; p = 0.05, ANOVA; degrees of freedom for medication group = 2 (group)

ADVERSE EVENTS:
Arm/Group | Placebo Group | Active Group: Sertraline Alone | Active Group: Sertraline Plus Gabapentin
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/36 | 1/30
Other Adverse Events (participants affected / at risk) | 7/36 | 17/36 | 14/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=36) | Active Group: Sertraline Alone (N=36) | Active Group: Sertraline Plus Gabapentin (N=30)
Allergic Reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) — Allergic reaction to study medication
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Group (N=36) | Active Group: Sertraline Alone (N=36) | Active Group: Sertraline Plus Gabapentin (N=30)
sexual dysfunction (Reproductive system and breast disorders) | 1 (1) | 4 (4) | 0 (0) — erectile dysfunction/impotence/inability or delayed orgasm
Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) — Chest pain in which cardiac involvement was ruled out.
dizziness (Cardiac disorders) | 2 (2) | 0 (0) | 1 (3) — self-reported dizziness
headache (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2)
Nausea and/or Emesis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 5 (7)
High Blood Pressure (Cardiac disorders) | 2 (3) | 3 (3) | 2 (3)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
toothache and/or tooth abscess (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 4 (4)
Skin Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2)
Anxiety (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Sore Throat (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Yawning (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No